CLINICAL TRIAL: NCT04655183
Title: A Phase I Dose Escalation Study of ATR Inhibitor M4344 in Combination With Niraparib in Participants With Advanced Solid Tumors Followed by Phase II Cohort Expansion in Participants With Breast Cancer With DNA Damage Response (DDR) Mutations
Brief Title: Study of M4344 in Combination With Niraparib
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Trial withdrawn based on portfolio prioritization; oral ATRi M1774 in combination with niraparib is under investigation in DDRiver Solid Tumor 301
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS201922_0010
Record Dates: First submitted 2020-11-27; First posted 2020-12-07 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Advanced Solid Tumor; Breast Cancer
Keywords: M4344; MSC2580591A; VX-803; VRT 1228692; ATR inhibitor; Advanced Solid Tumor; Breast Cancer; Niraparib
MeSH Terms: conditions — Breast Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1A (Dose escalation): Niraparib plus M4344 once daily (Experimental): Participants with baseline body weight < 77 kilograms (kg) or baseline platelet count < 150, 000 per cubic millimeter will be included in this Part. Dose escalation of M4344 administered along with niraparib.
  Interventions: Drug: Niraparib; Drug: M4344
- Part 1B (Dose escalation): Niraparib plus M4344 once daily (Experimental): Participants with baseline body weight > =77 kilograms (kg) and baseline platelet count >=150, 000 per cubic millimeter will be included in this Part. M4344 will be administered at a dose and schedule that was determined as the recommended dose for expansion (RDE) in Part 1A. Dose of niraparib will be escalated to the next higher dose level.
  Interventions: Drug: M4344; Drug: Niraparib
- Part 2 (Dose expansion): PARPi resistant, Niraparib plus M4344 (Experimental): Participants with Poly(ADP-ribose) polymerase inhibitor (PARPi) resistant, germline breast cancer 1/2 mutated (gBRCA1/2m) human epidermal growth factor receptor 2 (HER2) negative advanced Breast Cancer (aBC) will receive the combination of niraparib and M4344 at the RDE which was determined in Part 1.
  Interventions: Drug: Niraparib; Drug: M4344
- Part 3 (Dose expansion): PARPi-naive, Niraparib (Experimental): Participants with PARPi-naive germline BRCA1/2 wild type (gBRCAwt) homologous recombination repair gene mutated (HRRm) advanced breast cancer (aBC) will be randomized to receive niraparib as a single agent.
  Interventions: Drug: Niraparib
- Part 3 (Dose expansion): PARPi-naive, Niraparib plus M4344 (Experimental): Participants with PARPi-naive germline BRCA1/2 wild type (gBRCAwt) homologous recombination repair gene mutated (HRRm) advanced breast cancer (aBC) will be randomized to receive the combination of niraparib and M4344 at the RDE as determined in Part 1 of this study.
  Interventions: Drug: Niraparib; Drug: M4344

INTERVENTIONS:
Drug: Niraparib — Niraparib will be administered orally, once daily.
  Arms: Part 1A (Dose escalation): Niraparib plus M4344 once daily
Drug: M4344 — M4344 will be administered once daily or on an intermittent schedule in combination with niraparib.
  Other Names: MSC2580591A; VRT 1228692; VX-803
  Arms: Part 1A (Dose escalation): Niraparib plus M4344 once daily
Drug: Niraparib — Niraparib will be administered orally once daily at the RDE as determined in Part 1 of this study.
  Arms: Part 2 (Dose expansion): PARPi resistant, Niraparib plus M4344; Part 3 (Dose expansion): PARPi-naive, Niraparib plus M4344
Drug: M4344 — M4344 will be administered at a dose and schedule that was determined as RDE in Part 1A in combination with niraparib.
  Other Names: MSC2580591A; VRT 1228692; VX-803
  Arms: Part 1B (Dose escalation): Niraparib plus M4344 once daily; Part 2 (Dose expansion): PARPi resistant, Niraparib plus M4344; Part 3 (Dose expansion): PARPi-naive, Niraparib plus M4344
Drug: Niraparib — Niraparib will be administered orally, once daily. Dose of niraparib will be escalated beyond the dose in Part 1A.
  Arms: Part 1B (Dose escalation): Niraparib plus M4344 once daily
Drug: Niraparib — Niraparib will be administered as single agent at the approved dose.
  Arms: Part 3 (Dose expansion): PARPi-naive, Niraparib

SUMMARY:
Study will include 3 parts. Aim of Part 1 of this study is to establish the maximum tolerated dose (MTD) and recommended dose for expansion (RDE) for M4344 (is an Ataxia Telangiectasia Mutated and Rad3-related [ATR] inhibitors) in combination with niraparib in participants with advanced solid tumors. Aim of Parts 2 and 3 of the study is to provide clinical proof-of-concept for the preclinically predicted synergistic efficacy of ATR and poly(ADP-Ribose) polymerase (PARP) inhibitors (PARPi) in defined populations of participants with advanced breast cancer (aBC) with DDR mutations with an unmet medical need.

ELIGIBILITY:
Inclusion Criteria:

* Participants in All Parts:
* Have Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1 (ECOG 0-2 for Phase II)
* Participants with human immunodeficiency virus (HIV) infection are eligible if they are on effective anti-retroviral therapy with undetectable viral load within 6 months, provided there is no expected drug-drug interaction
* Participants with a history of hepatitis C virus (HCV) infection are eligible if they have been treated and cured
* Participants in Part 1:
* Are participants with advanced solid tumors, except for advanced prostate cancer, for whom no standard of care therapy exists, or in whom conventional therapy is not reliably effective, or in whom treatment with study intervention can be reasonably expected to provide clinical benefit
* Participants in Part 2:
* Are participants with advanced Germline Breast Cancer Gene (BRCA)1/2-Mutant Wild Type (gBRCA1/2)-mutant, Poly(ADP-Ribose) Polymerase Inhibitor(s) (PARPi)-resistant Human Epidermal Growth Factor Receptor 2 Negative (HER2)- breast cancer. There is no limit for prior lines of chemotherapy for metastatic disease
* Participants with at least one measurable lesion that is suitable for repeated assessment as per RECIST 1.1
* Participants in Part 3:
* Are participants with advanced BRCA1/2 wild-type, Homologous Recombination Repair Gene Mutated (HRRm) Human Epidermal Growth Factor Receptor 2 Negative (HER2)- breast cancer
* Participants must not have had prior treatment with a PARPi in any disease setting
* All participants with at least one measurable or non-measurable but evaluable lesion that is suitable for repeated assessment as per RECIST 1.1
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with clinically relevant (that is [i.e], active), uncontrolled intercurrent illness including, but not limited to, severe active infection (i.e. requiring hospitalization and/or intravenous antibiotics), uncontrolled arterial hypertension, i.e. systolic blood pressure (BP) > 140 millimeter of mercury (mmHg), diastolic BP > 90 mmHg, symptomatic congestive heart failure (>= New York Heart Association Classification Class II), unstable angina pectoris or myocardial infarction, cardiac arrhythmia requiring medication, cerebral vascular accident/stroke, or any psychiatric illness/social situations that would limit compliance with study requirements
* Participants with a known additional malignancy that is progressing and/or requires active treatment. In addition, participants must not have a known history or current diagnosis of Myelodysplastic Syndrome (MDS) or Acute Myeloid Leukemia (AML) at any time or have been diagnosed with another malignancy within 3 years of starting treatment. Exceptions include fully resected basal cell carcinoma of the skin or squamous cell carcinoma of the skin, in situ cervical cancer, fully resected ductal carcinoma in situ, and Stage IA, Grade I endometrioid endometrial cancer with no myometrial invasion, that has undergone curative therapy
* Participants diagnosed with hereditary diseases characterized by genetic defects of Deoxyribonucleic acid (DNA) repair mechanisms, including ataxia telangiectasia, Nijmegen breakage syndrome, Werner syndrome, Bloom Syndrome, Fanconi anemia, xeroderma pigmentosum, Cockayne syndrome, and trichothiodystrophy
* Treatment with live or live attenuated vaccine within 30 days of dosing
* Participants with clinically relevant, uncontrolled intercurrent illness, unstable brain metastases, has a known additional malignancy that is progressing and/or requires active treatment
* Received hematopoietic growth factor (example, granulocyte colony-stimulating factor, erythropoietin) within 14 days prior to the first dose of study intervention
* Participants receiving treatment with proton-pump inhibitors that cannot be discontinued at least 1 week before first dose of study intervention and for the duration of the study
* Other protocol defined inclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Part 1 A and B: Number of Participants with Dose Limiting Toxicities (DLTs) | Day 1 up to Day 28
Part 1 A and B: Number of Participants with Treatment Emergent Adverse Events (TEAEs), Serious TEAEs and Treatment-related TEAEs | From Baseline until 6.5 months
Part 2: Objective response (OR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 Assessed by Investigator | From Baseline until disease progression (assessed up to approximately 1 years)
Part 3: Progression Free Survival (PFS) According to RECIST Version 1.1 Assessed by Investigator | From Baseline until disease progression or death (assessed up to approximately 1 years)

SECONDARY OUTCOMES:
Part 1 A and B: Number of Participants with Clinically Significant Changes From Baseline in Vital Signs, 12-Lead Electrocardiogram (ECG) Assessments Findings and Laboratory parameters | From Baseline until 6.5 months
  Number of participants with clinically significant changes from baseline in vital signs, 12-Lead Electrocardiogram (ECG) assessments findings and laboratory parameters will be reported.
Part 1A and B: Objective response (OR) According to RECIST Version 1.1 Assessed by Investigator | From Baseline until disease progression (assessed up to approximately 6.5 months)
Part 1 A and B: Area Under the Concentration-time Curve From Time Zero to the Last Sampling time (AUC 0-tlast) of M4344, Metabolites of M4344 and Niraparib | Cycle 1 Day 1 to Cycle 4 Day 1 and every second cycle thereafter Day 1 (each cycle is of 28 days), assessed up to approximately 6.5 months
Part 1A and B: Area Under Plasma Concentration-Time Curve Within One Dosing Interval (AUC0-tau) of M4344, Metabolites of M4344 and Niraparib | Cycle 1 Day 1 to Cycle 4 Day 1 and every second cycle thereafter Day 1 (each cycle is of 28 days), assessed up to approximately 6.5 months
Part 1A and B: Dose Normalized Area Under Concentration-Time Curve Within One Dosing Interval (AUC0-tau/Dose) of M4344, Metabolites of M4344 and Niraparib | Cycle 1 Day 1 to Cycle 4 Day 1 and every second cycle thereafter Day 1 (each cycle is of 28 days), assessed up to approximately 6.5 months
Part 1A and B: Dose Normalized Area Under Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC0-last/Dose) of M4344, Metabolites of M4344 and Niraparib | Cycle 1 Day 1 to Cycle 4 Day 1 and every second cycle thereafter Day 1 (each cycle is of 28 days), assessed up to approximately 6.5 months
Part 1A and B: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of M4344, Metabolites of M4344 and Niraparib | Cycle 1 Day 1 to Cycle 4 Day 1 and every second cycle thereafter Day 1 (each cycle is of 28 days), assessed up to approximately 6.5 months
Part 1A and B: Dose Normalized Area Under Concentration-Time Curve From Time Zero (dosing time) Extrapolated to Infinity (AUC0-inf/Dose) of M4344, Metabolites of M4344 and Niraparib | Cycle 1 Day 1 to Cycle 4 Day 1 and every second cycle thereafter Day 1 (each cycle is of 28 days), assessed up to approximately 6.5 months
Part 1A and B: Area Under Concentration From Time tlast Extrapolated to Infinity (AUCextra%) of M4344, Metabolites of M4344 and Niraparib | Cycle 1 Day 1 to Cycle 4 Day 1 and every second cycle thereafter Day 1 (each cycle is of 28 days), assessed up to approximately 6.5 months
Part 1A and B: Apparent Total Body Clearance From Plasma (CL/f) of M4344, Metabolites of M4344 and Niraparib | Cycle 1 Day 1 to Cycle 4 Day 1 and every second cycle thereafter Day 1 (each cycle is of 28 days), assessed up to approximately 6.5 months
Part 1A and B: Apparent Total Body Clearance From Plasma at Steady State Following Extravascular Administration (CLss/F) of M4344, Metabolites of M4344 and Niraparib | Cycle 1 Day 1 to Cycle 4 Day 1 and every second cycle thereafter Day 1 (each cycle is of 28 days), assessed up to approximately 6.5 months
Part 1A and B: Maximum Observed Concentration (Cmax) of M4344, Metabolites of M4344 and Niraparib | Cycle 1 Day 1 to Cycle 4 Day 1 and every second cycle thereafter Day 1 (each cycle is of 28 days), assessed up to approximately 6.5 months
Part 1A and B: Dose Normalized Maximum Observed Concentration (Cmax/Dose) of M4344, Metabolites of M4344 and Niraparib | Cycle 1 Day 1 to Cycle 4 Day 1 and every second cycle thereafter Day 1 (each cycle is of 28 days), assessed up to approximately 6.5 months
Part 1A and B: Plasma Concentration Observed Immediately Before Next Dosing (Ctrough) of M4344, Metabolites of M4344 and Niraparib | Cycle 1 Day 1 to Cycle 4 Day 1 and every second cycle thereafter Day 1 (each cycle is of 28 days), assessed up to approximately 6.5 months
Part 1A and B: Metabolic Ratio of Area Under Plasma Concentration-Time Curve Within One Dosing Interval MR(AUC0-tau) of M4344, Metabolites of M4344 and Niraparib | Cycle 1 Day 1 to Cycle 4 Day 1 and every second cycle thereafter Day 1 (each cycle is of 28 days), assessed up to approximately 6.5 months
Part 1A and B: Metabolic Ratio of Maximum Observed Concentration MR(Cmax) of M4344, Metabolites of M4344 and Niraparib | Cycle 1 Day 1 to Cycle 4 Day 1 and every second cycle thereafter Day 1 (each cycle is of 28 days), assessed up to approximately 6.5 months
Part 1A and B: Accumulation Ratio for AUCtau (Racc[AUCtau]) of M4344, Metabolites of M4344 and Niraparib | Cycle 1 Day 1 to Cycle 4 Day 1 and every second cycle thereafter Day 1 (each cycle is of 28 days), assessed up to approximately 6.5 months
Part 1A and B: Accumulation Ratio for Maximum Observed Concentration (Racc[Cmax]) of M4344, Metabolites of M4344 and Niraparib | Cycle 1 Day 1 to Cycle 4 Day 1 and every second cycle thereafter Day 1 (each cycle is of 28 days), assessed up to approximately 6.5 months
Part 1A and B: Apparent Terminal Half-life (t1/2) of M4344, Metabolites of M4344 and Niraparib | Cycle 1 Day 1 to Cycle 4 Day 1 and every second cycle thereafter Day 1 (each cycle is of 28 days), assessed up to approximately 6.5 months
Part 1A and B: Time to Reach Maximum Plasma Concentration (tmax) of M4344, Metabolites of M4344 and Niraparib | Cycle 1 Day 1 to Cycle 4 Day 1 and every second cycle thereafter Day 1 (each cycle is of 28 days), assessed up to approximately 6.5 months
Part 1A and B: Apparent Volume of Distribution During Terminal Phase Following Extravascular Administration (Vz/F) of M4344, Metabolites of M4344 and Niraparib | Cycle 1 Day 1 to Cycle 4 Day 1 and every second cycle thereafter Day 1 (each cycle is of 28 days), assessed up to approximately 6.5 months
Part 2 and Part 3: Number of Participants with Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, and Treatment-related TEAEs | From Baseline and up to 1 year
  Number of participants with clinically significant changes from baseline in vital signs, 12-Lead Electrocardiogram (ECG) assessments findings and laboratory parameters will be reported.
Part 2 and Part 3: Number of Participants with Clinically Significant Change From Baseline in Vital Signs, 12-Lead Electrocardiogram (ECG) Assessments Findings and Laboratory parameters | From Baseline up to 1 year
Part 2: Progression Free Survival (PFS) According to RECIST Version 1.1 Assessed by Investigator | From Baseline until disease progression or death (assessed up to approximately 1 years)
Part 2 and Part 3: Overall Survival (OS) | From Baseline until study closure or death, whichever comes first (assessed up to approximately 1 years)
Part 2 and Part 3: Duration of Response (DOR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | From Baseline until disease progression or death (assessed up to approximately 1 years)
Part 3:Objective response (OR) According to RECIST Version 1.1 Assessed by Investigator | From Baseline until disease progression (assessed up to approximately 1 years)
Part 2 and Part 3: Concentrations of M4344, Metabolites of M4344 and Niraparib | Cycle 1, Day 1 to Cycle 2 Day 1 and subsequently every other cycle Day 1 (each cycle is of 28 days), assessed up to approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany

IPD SHARING:
Plan to Share IPD: Yes
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, EMD Serono will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.emdgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html